CLINICAL TRIAL: NCT05247177
Title: Effects of Multimodal General Anesthesia for Older Patients Undergoing Lumbar Spine Fusion Surgery: a Randomized Controlled Trial
Brief Title: Multimodal GA for Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202112040MIND
Record Dates: First submitted 2022-02-06; First posted 2022-02-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Spine Fusion Surgery
Keywords: multimodal general anesthesia,lumbar spine surgery,electroencephalographic,EEG,density spectrum array,DSA,bispectral index(BIS)
MeSH Terms: interventions — Dexmedetomidine; Sevoflurane; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal general anesthesia (Experimental): General anesthesia maintained by co-administration of sevoflurane, dexmedetomidine and ketamine by using a predefined EEG density spectrum array pattern
  Interventions: Drug: dexmedetomidine, ketamine co-administration with sevoflurane for general anesthesia
- Conventional general anesthesia (Active Comparator): General anesthesia maintained by administration of sevoflurane alone to keep a bispectral index between 40-60
  Interventions: Drug: Conventional general anesthesia by administration of sevoflurane alone

INTERVENTIONS:
Drug: dexmedetomidine, ketamine co-administration with sevoflurane for general anesthesia — co-administration of sevoflurane, iv. dexmedetomidine and iv. ketamine to maintain a predefined EEG density spectrum array pattern for general anesthesia
  Arms: Multimodal general anesthesia
Drug: Conventional general anesthesia by administration of sevoflurane alone — Administration of sevoflurane alone to maintain anesthesia with a bispectral index between 40-60
  Arms: Conventional general anesthesia

SUMMARY:
To evaluate the effects of multimodal general anesthesia on the recovery profile of elder patients undergoing lumbar spine fusion surgery.

DETAILED DESCRIPTION:
Multimodal general anesthesia has been proposed in recent years. By administration of multiple agents acting on a different component of the nociceptive pathways, the multimodal general anesthesia may elicit maximal anesthetic effects with minimal anesthetic dose. These may be beneficial to improve postoperative recovery and reduce adverse effects such as postoperative delirium and perioperative neurocognitive impairment. It is not uncommon that elder patients undergoing lumbar spine fusion surgery suffer from postoperative poor recovery, postoperative delirium as well as the postoperative neurocognitive disorder. Therefore, this study aims to explore the potential effects of multimodal general anesthesia, which comprised with electroencephalography density spectrum array guided co-administration of sevoflurane, ketamine and dexmedetomidine, on the postoperative recovery profiles for elder patients undergoing lumbar spine fusion surgery.

ELIGIBILITY:
Inclusion criteria:

1. patients with ages at least 60-year undergoing elective lumbar spine surgery

Exclusion:

1. A history of dementia
2. Impaired liver function, eg. AST or ALT >100; liver cirrhosis > Child B class
3. Impaired renal function, cGFR< 60 ml/min/1.73 m2
4. Cardiac dysfunction, such as heart failure > NYHA class II

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Quality of Recovery Score | Change from Baseline QoR-15 to 24 hour after surgery
  Postoperative Quality of Recovery Score assessed by using the QoR-15 system

SECONDARY OUTCOMES:
Postoperative delirium | 3 days
  Postoperative delirium assessed by using the confusion assessment method (CAM) daily at least once for 3 days
Postoperative chronic pain | 3 months
  Postoperative chronic pain intensity at 3 months after surgery assessed by using the Brief Pain Inventory questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan